CLINICAL TRIAL: NCT02767453
Title: The Utility of Closed Suction Drainage in Total Shoulder Arthroplasty: A Prospective Analysis.
Brief Title: Closed Suction Drainage in Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Christopher S. Ahmad, MD, Professor of Orthopedic Surgery at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAO2805
Record Dates: First submitted 2016-05-04; First posted 2016-05-10 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis
Keywords: Shoulder arthroplasty; Closed suction drainage; Glenohumeral; Drainage tube
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Shoulder; theasinensin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TSA with drain placement (Active Comparator): Hemovac drains are placed in subjects during standard Total Shoulder Arthroplasty involving the replacement of damaged shoulder components with shoulder prosthesis.
  Interventions: Procedure: Wound drainage; Procedure: Total Shoulder Arthroplasty
- TSA without drain placement (Active Comparator): Hemovac drains will not be placed in subjects during standard Total Shoulder Arthroplasty involving the replacement of damaged shoulder components with shoulder prosthesis.
  Interventions: Procedure: Total Shoulder Arthroplasty

INTERVENTIONS:
Procedure: Wound drainage — Experimental portion removing/draining blood/fluid from a space created during a surgical procedure. Typically, surgeons place a plastic tube in the shoulder joint to drain fluids that may accumulate after surgery. Hemovac drain is a FDA-approved device routinely used or wound drainage; however, there is no known evidence whether this improves outcomes of surgery.
  Arms: TSA with drain placement
Procedure: Total Shoulder Arthroplasty — Standard procedure for treating the severe pain and stiffness that often result at the end stage of various forms of arthritis or degenerative joint disease of the shoulder joint. The primary goal of shoulder replacement surgery is pain relief, with a secondary benefit of restoring motion, strength, function, and assisting with returning patients to an activity level as near to normal as possible. Shoulder prosthesis is a standard artificial device to replace both components of the "ball and socket" joint during TSA.
  Other Names: TSA

SUMMARY:
The purpose of this study is to determine the limited effectiveness of drains during Total Shoulder Arthroplasty. Drains are used during joint arthroplasty procedures to decrease infection rates, swelling,and the number of dressing changes required during a hospital stay. The use of drains has been heavily investigated in the hip and knee replacement literature, but there have been no investigations regarding their use in shoulder replacements, despite frequent use.

Clinical benefit has not been consistently documented regarding drain usage in hip and knee arthroplasty and the investigators hypothesize that they are of limited utility in total shoulder arthroplasty as well. The investigators will perform a prospective investigation of total shoulder arthroplasty patients- dividing them into two groups- half will receive a drain at the time of surgery and the other half will not be receiving a drain.

DETAILED DESCRIPTION:
The use of closed-suction draining has been well studied in the hip and knee arthroplasty literature. Drains have been used with the intention of decreasing infection, ecchymoses, and frequency of dressing changes. Some have reported a corresponding decrease in hematocrit for patients receiving post-op drainage leading to increased transfusion needs. Given that no clinical benefit has been consistently documented regarding drain usage in knee and hip arthroplasty, they are no longer routinely used in those operations. The use of such drainage systems in shoulder arthroplasty, however, has not been studied and the benefit of drain use in regards to patient outcomes is questionable. As such, the study is a prospective investigation comparing outcomes in two groups of total shoulder arthroplasty patients, those receiving a drain at the time of surgery and those without a drain. The short-term outcome measurements include peri-operative hematocrit and hemoglobin, infection rate, hematoma development, transfusion requirement, ecchymosis and wound complication. Long-term outcomes include shoulder functional scores as measured by post-operative visits and any need for revision shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Glenohumeral Osteoarthritis undergoing total shoulder arthroplasty

Exclusion Criteria:

* Patients undergoing total shoulder arthroplasty following trauma, failed prior surgery/revision or infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin level | Day 0 post-operative, day 1 post-operative, day 2 post-operative
  To assess blood loss
Change in Hematocrit level | Day 0 post-operative, day 1 post-operative, day 2 post-operative
  To assess blood loss

SECONDARY OUTCOMES:
Total length of hospital stay | Day 0 post-operative to discharge, an average of up to 3 days
  Calculated in number of days
Total cost incurred during hospital stay | Pre-surgical admitting to discharge, an average of up to 3 days
  Calculation will include the cost of the surgical procedure
Change in Elbow Surgeons Evaluation Form (ASES) score | Baseline, 6 month post-operative, 1 year post-operative, 2 year post-operative
  To determine the longterm effect of drain usage on functional shoulder score-total score from 0-100 where 0= worse pain and functional loss /disability
Number of subjects that developed any of the following: wound compromise, ecchymosis, bleeding, hematoma formation or infection | Day 0 post-operative to discharge, an average of up to 3 days
Total Drain Output record | Day 1 post-operative, day 2 post-operative
  Calculated total blood loss in ml
Number of subjects that presented with anatomic healing after total shoulder arthroplasty | 6 month post-operative, 1 year post-operative, 2 year post-operative
  To be determined by shoulder ultrasound results
Change in Disabilities of the Arm Shoulder and Hand (DASH) Score | Baseline, 6 month post-operative, 1 year post-operative, 2 year post-operative
  To determine the longterm effect of drain usage on functional shoulder score- measured from 0-100 a higher score indicates greater disability

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S. Ahmad, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No